CLINICAL TRIAL: NCT06990984
Title: A Phase 2a Partially Randomized, Placebo-controlled, Sequential Dose-ranging Study of TTI-0102 in Adults and Children With Leigh Syndrome Spectrum
Brief Title: A Dose-ranging Study of TTI-0102 in Adults and Children With Leigh Syndrome Spectrum (LSS)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thiogenesis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTI-LSS-001
Record Dates: First submitted 2025-05-06; First posted 2025-05-25 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Leigh Syndrome
MeSH Terms: conditions — Leigh Disease | interventions — cysteamine-pantetheine disulfide; Mannitol

STUDY DESIGN:
Intervention Model Description: partially randomized, placebo-controlled, sequential dose-ranging treatment study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties will be blinded during the placebo-controlled Sequence 1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TTI-0102: cysteamine-pantetheine disulfide (Experimental)
  Interventions: Drug: TTI-0102: cysteamine-pantetheine disulfide
- Placebo (Placebo Comparator)
  Interventions: Drug: D-Mannitol

INTERVENTIONS:
Drug: TTI-0102: cysteamine-pantetheine disulfide — TTI-0102: cysteamine-pantetheine disulfide, powder for dissolution in water for oral administration
  Arms: TTI-0102: cysteamine-pantetheine disulfide
Drug: D-Mannitol — D-Mannitol
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate oral TTI-0102 to evaluate its pharmacokinetics, safety, and preliminary efficacy in patients with Leigh syndrome spectrum, in three sequences. First sequence will be placebo-controlled and include 12 adolescents and adults weighing more than 40 kg. Second sequence will be open-label and include 3 adults and 3 children weighing 25-40 kg. Third sequence will also be open-label and will include 3 children weighing 20-25 kg. The main questions clinical trial aims to answer are:

* Characterize the relationship between TTI-0102 drug levels by measuring

  1. cysteamine pharmacokinetic (PK) parameters
  2. pharmacodynamic (PD) efficacy measures
* Generate a population PK model and determine dose level for later dosing groups
* collect data to inform the design of a subsequent phase 2b/3 study of TTI-0102 in this patient population

Participants will be asked to:

* Take the study drug twice daily for 12 weeks
* Visit the clinic for checkups and testing 7 times in total: once prior to study drug dosing, then 5 times over the 12-week treatment period and one more time a month after the last study drug dose.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 5 years to 55 years (inclusive) and weight-eligible, at the time of informed consent / assent and enrollment
* Confirmed diagnosis of Leigh syndrome or Leigh-like disorder (Leigh syndrome spectrum [LSS]) with neurodevelopmental manifestations, which include documented developmental delay, developmental regression, or abnormal neurologic exam findings
* Willing and able to comply with required study schedule and procedures, including daily TTI-0102 study drug dosing requirements, i.e., able to ingest solution orally
* Adequate liver function as evidenced by total bilirubin < 1.5x upper limit of normal (ULN) and liver function tests < 3x ULN
* Normal hematologic parameters defined as:

Absolute neutrophil count ≥ 1.0 x 109/L Platelet count ≥ 100,000/mm3 (100 x 109/L) Hemoglobin ≥ 9 g/dL

* Non-fasting serum triglycerides < 300 mg/dL and non-fasting serum cholesterol < 300 mg/dL
* Serum amylase and lipase < 2x ULN
* Adequate immunoglobulin levels as outlined below that, in the opinion of the investigator, will not place the patient at increased risk of infection:

IgG ≥ 200 mg/dL IgM ≥ 30 mg/dL IgA ≥ 10 mg/dL

* All sexually-active participants must agree to use effective contraception during study participation:

  1. Females of reproductive potential must agree to use effective contraception without interruption from 28 days prior to starting TTI-0102 through 30 days after last dose of TTI-0102; have a negative serum pregnancy test result at screening; and agree to ongoing urine pregnancy testing during the subsequent study period.
  2. Male patients must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of reproductive potential while participating in the study and through 30 days after the last dose of TTI-0102

     Exclusion Criteria:
* Documented diagnosis of concurrent inborn errors of metabolism
* Non-elective hospitalization related to their Leigh syndrome or mitochondrial disease within 60 days prior to screening
* Treatment with taurine during the previous 30 days of screening, and not willing to discontinue for the duration of the study
* Severe gastrointestinal disease including gastroparesis
* Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* In the opinion of the investigator, clinically-significant or severe cardiac conditions, at the time of screening
* History of drug or alcohol abuse
* History of pancreatitis
* Known or suspected hypersensitivity to cysteamine
* Allergy to any medicine containing mercaptamine, penicillamine, or known hypersensitivity to any of the study drug ingredients
* Exposure to any live vaccinations within 30 days prior to the first dose of TTI-0102, except for the influenza and / or COVID-19 vaccines
* Planned surgical procedure during the study period
* Clinically-significant proteinuria that requires ongoing medical therapy
* Patients who are breastfeeding and / or are pregnant
* History of solid organ transplant or bone marrow transplant
* Treatment with any investigational drug, including an investigational drug for mitochondrial disease, within 30 days prior to receiving the first dose of TTI-0102
* Patients with confirmed or suspected increased intracranial pressure, pseudotumor cerebri / idiopathic intracranial hypertension, and or papilledema
* Currently active malignancy (other than adequately treated non-melanoma skin cancers, carcinoma in situ of the cervix, or other adequately treated carcinoma in situ) and / or ongoing treatment for malignancy are ineligible. Patients are not considered to have a currently active malignancy if they have completed therapy and are free of disease for at least one year
* Recent infection requiring systemic anti-infective treatment that was completed ≤ 14 days prior to screening
* Uncontrolled diabetes mellitus, as defined by HbA1c > 8%, despite adequate therapy
* History of interstitial lung disease and / or pneumonitis
* Known human immunodeficiency virus, active hepatitis B and / or hepatitis C infection(s)
* Any uncontrolled psychiatric or medical condition which, in the opinion of the investigator, would interfere with the patient's safe participation in the study
* Any other condition or prior therapy that in the opinion of the investigator would render the participant unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol and / or likelihood of non-compliance with any study requirements

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
PK: plasma cysteamine (Tmax) | Baseline (Day 1) to end of treatment (Day 84)
  Measurement of cysteamine in plasma: Tmax
PK: plasma cysteamine (Cmax) | Baseline (Day 1) to end of treatment (Day 84)
  Measurement of cysteamine in plasma: Cmax
PK: plasma cysteamine (Cmin) | Baseline (Day 1) to end of treatment (Day 84)
  Measurement of cysteamine in plasma: Cmin
PK: plasma cysteamine (PK curve) | Baseline (Day 1) to end of treatment (Day 84)
  Measurement of cysteamine in plasma: PK curve
PK: plasma cysteamine (AUC) | Baseline (Day 1) to end of treatment (Day 84)
  Measurement of cysteamine in plasma: AUC
PD: plasma glutathione | Baseline (Day 1) to end of treatment (Day 84)
  Measurement of glutathione concentration in plasma

SECONDARY OUTCOMES:
Safety and adverse events | Baseline (Day 1) to final follow-up (Day 112)
  Number of participants with treatment-emergent adverse events [comparing active vs. placebo]

CONTACTS AND LOCATIONS:
Overall Officials: Zarazuela Zolkipli-Cunningham, MBChB, MRCP, Principal Investigator — Children's Hospital of Philadelphia; Patrice Rioux, MD, PhD, Study Director — Thiogenesis Therapeutics

IPD SHARING:
Plan to Share IPD: Undecided
This is an exploratory study and we are not certain yet what data will be shared with other researchers.